CLINICAL TRIAL: NCT00296218
Title: Randomized Comparison of a Two-month Regimen of Irbesartan Versus Enalapril on Cardiovascular Markers in Patients With Acute Coronary Syndrome Without ST Segment Elevation.
Brief Title: ARCHIPELAGO: Irbesartan in Patients With Acute Coronary Syndrome Without ST Segment Elevation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PM_C_0024; EudraCT #: 2005-002161-36
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Myocardial Ischemia; Hypertension
MeSH Terms: conditions — Myocardial Ischemia; Hypertension | interventions — Irbesartan

INTERVENTIONS:
Drug: Irbesartan

SUMMARY:
Primary Objective

* The main objective of this study is to assess if a two-month regimen of irbesartan in patients hospitalized for acute coronary syndrome without ST segment elevation can reduce inflammation markers (ie hsCRP), in comparison to a similar regimen of enalapril.

Secondary Objectives

* To compare both regimens on several other biological parameters which have demonstrated their relevance and their predictive clinical value (ie BNP, microalbuminuria, troponin I …) in this patient population.
* To compare on the above parameters the early initiation of treatment versus the initiation of treatment at hospital discharge.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria

* Patient hospitalised with ischemic symptoms (last episode within the last 48 hours before randomization) and at least one of the following characteristics of NSTEACS (non-ST-segment-elevation acute coronary syndromes):

  * ECG ST or T changes (ST depression or transient elevation of at least 1mm or T wave changes in at least 2 leads)
  * Positive troponin (according to local threshold)

Exclusion Criteria

* Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study WOCBP using a prohibited contraceptive method (not applicable)
* Women who are pregnant or breast feeding
* Women with a positive pregnancy test on enrolment or prior to study drug administration
* Patient with dementia
* Persistent ST segment elevation at ECG
* Systolic blood pressure < 100 mmHg
* Bilateral stenosis of renal artery
* Creatinine clearance < or = 30ml/mn
* Congestive heart failure with symptoms consistent with New York Heart Association (NYHA) class III or IV.
* Aortic or mitral valve stenosis
* Hypertrophic cardiomyopathy
* Connective tissue disease with vascular involvement
* Angioplasty, surgery or trauma within the last 3 months
* Coronarography or angioplasty planned to be performed or performed before baseline sampling
* Febrile (≥ 38°C) disease, known concomitant viral or bacterial infection, chronic auto immune disease, chronic inflammatory disease, known cancer in evolution
* Hyperkalemia: serum potassium > 5.5mmol/l
* Sensitivity or intolerance to Angiotensin receptor blockers (ARBs) : olmesartan, candesartan, irbesartan, eprosartan, losartan, telmisartan, valsartan and/or any other ARB currently or previously in development.
* Sensitivity or intolerance to Angiotensin-converting Enzyme Inhibitors (ACE-I) : benazepril, captopril, enalapril, lisinopril, trandolapril, ramipril, quinapril, and/or any other ACE-I currently or previously in development.
* Chronic steroid or non-steroidal anti inflammatory drugs (NSAIDs) use. Aspirin is permitted.
* Treatment with allopurinol or procaïnamide
* Concomitant use of potassium sparing diuretics (eg. spironolactone, triamterene or amiloride), potassium preparations or salt substitutes containing potassium
* Treatment with Lithium
* Immunosupressive medication
* Administration of any other investigational drug in the last 30 days before enrolment and during the course of the study
* Treatment with ARB or ACE inhibitor within the last 3 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2006-02; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
comparison of the relative change from baseline in hsCRP at day 60 between the two treatment groups

SECONDARY OUTCOMES:
Relative change from baseline of hsCRP at discharge
Changes from baseline in BNP and Microalbuminuria (MAU) at discharge and day 60
Change of Troponin I from baseline at discharge
In addition at baseline, discharge and D60 the following parameters will be evaluated and their evolution compared in the two treatment groups: IL6, CD 40 L, sPLA2 and Lp-PLA2, IMA, MMP-9, MPO (myeloperoxydase), aldosterone
Blood pressure at discharge, D15 and D60.
The early versus late (at hospital discharge) initiation of treatment will also be evaluated on the above-listed parameters.
& Safety outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Domenger, MD, Study Director — Sanofi
Locations (11):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Meyrin, Switzerland
- Sanofi-Aventis, Guildford, United Kingdom

REFERENCES:
- [Result] Montalescot G, Drexler H, Gallo R, Pearson T, Thoenes M, Bhatt DL. Effect of irbesartan and enalapril in non-ST elevation acute coronary syndrome: results of the randomized, double-blind ARCHIPELAGO study. Eur Heart J. 2009 Nov;30(22):2733-41. doi: 10.1093/eurheartj/ehp301. Epub 2009 Aug 21. PMID 19700470